CLINICAL TRIAL: NCT06359756
Title: Ischemic Postconditioning in Prevention of Brain Damage After Carotid Surgery - a Clinical Trial for Vascular Evaluation
Brief Title: Ischemic Postconditioning in Carotid Surgery
Acronym: BRAIN-SAVE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Cardiovascular Diseases Dedinje (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BRAIN-SAVE1
Record Dates: First submitted 2024-04-06; First posted 2024-04-11 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Ischemic Postconditioning; Carotid Surgery; Stroke; Carotid Artery Diseases
Keywords: Ischemic Postconditioning; Carotid Surgery
MeSH Terms: conditions — Stroke; Carotid Artery Diseases | interventions — Ischemic Postconditioning

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ischemic postconditioning group (Experimental): Patients with ischemic postconditioning (IPCT) performed after standard eversion carotid endarterectomy (eCEA)
  Interventions: Procedure: Ischemic postconditioning in carotid surgery
- Control (Active Comparator): Patients with standard eversion carotid endarterectomy (eCEA) performed with no ischemic postconditioning (IPCT)
  Interventions: Procedure: Eversion Carotid Endarterectomy

INTERVENTIONS:
Procedure: Ischemic postconditioning in carotid surgery — After the initial declamping of the carotid artery the procedure is performed with 6 cycles of reperfusion of 30 seconds each (clamping of the internal carotid artery) which are successively followed by 6 cycles of ischemia lasting 30 seconds (clamping of the internal carotid artery). Clamping is done on the unaltered ICA, at the clamping site prior to performing CEA above the plaque termination point.
  Other Names: IPCT
  Arms: Ischemic postconditioning group
Procedure: Eversion Carotid Endarterectomy — Standard Eversion Carotid Endarterectomy
  Other Names: eCEA
  Arms: Control

SUMMARY:
Analyzing changes in cerebral oximetry, transcranial Doppler and biomarkers of neuronal ischemic injury and blood-brain barrier integrity assessing the safety and efficacy of ischemic postconditioning in carotid surgery (IPCT).

DETAILED DESCRIPTION:
Eversion carotid endarterectomy (eCEA) has proven effective in preventing ischemic brain damage resulting from atherosclerotic disease in the extracranial segment of the carotid arteries. Over time, advancements in surgical techniques have led to a reduction in the incidence of perioperative stroke. To better understand the concept of stroke complications following CEA, a clear distinction between intraprocedural and postprocedural strokes is necessary. Periprocedural strokes are attributed to hypoperfusion or embolization from the site of endarterectomy, while defined causes of postprocedural strokes include local carotid artery thrombosis or cerebral hyperperfusion syndrome (CHS).

CHS, occurring in 1-3% of cases, is a potentially catastrophic event following eCEA, primarily resulting from impaired autoregulation mechanisms and post-revascularization changes in cerebral hemodynamics. Patients with significant carotid stenosis are particularly vulnerable to CHS due to prolonged cerebral hypoperfusion, where collateral circulation serves as a protective mechanism. Another pathway leading to CHS involves increased free radical concentrations, damaging the blood-brain barrier. Identified risk factors for CHS development include advanced age, prior ischemic cerebrovascular events, and contralateral stenosis > 70%.

Various methods for predicting CHS development and collateral circulation insufficiency include cerebral oximetry, transcranial Doppler sonography, perfusion computed tomography, and quantitative magnetic resonance imaging. Cerebral oximetry, with real-time detection of cerebral oxygenated hemoglobin saturation, exhibits promising sensitivity and specificity in predicting CHS occurrence.

Analyzing changes in biomarkers of neuronal ischemic injury and blood-brain barrier integrity offers insight into CHS pathophysiology and indirectly assesses the safety and efficacy of ischemic postconditioning of the carotid artery (IPCT) in high-risk patients. IPCT, shown to have a protective effect in animal models, recently demonstrated encouraging results in human trials.

Utilizing intraoperative neuromonitoring with cerebral oximetry and transcranial Doppler enables real-time monitoring of cerebral oxygenated hemoglobin saturation and flow characteristics during and after IPCT, validating its protective effect and safety in high-risk CHS scenarios.

ELIGIBILITY:
Inclusion Criteria:

* unilateral carotid artery stenosis >90%
* bilateral stenosis >80%
* unilateral stenosis >80% with contralateral occlusion/subocclusion

Exclusion Criteria:

* urgent carotid endarterectomy
* carotid restenosis
* "major surgery" in the last 6 months
* malignant diseases
* previous brain trauma or surgery
* epilepsy

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with perioperative stroke | During and 30 days after surgery
Number of Participants with perioperative death | During and 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Nenad Ilijevski, PhD, Principal Investigator — Institute for Cardiovascular Diseases Dedinje
Locations (1):
- Institute for Cardiovascular Diseases Dedinje, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ilijevski N, Atanasijevic I, Lozuk B, Gajin P, Matic P, Babic S, Sagic D, Unic-Stojanovic D, Tanaskovic S. Direct Ischemic Postconditioning After Carotid Endarterectomy in the Prevention of Postoperative Cerebral Ischemic Complications-Observational Case-Control Study. J Cardiovasc Pharmacol Ther. 2022 Jan-Dec;27:10742484221137489. doi: 10.1177/10742484221137489. PMID 36377766